CLINICAL TRIAL: NCT03189030
Title: A Phase 1 Safety and Tolerability Study of Personalized Live, Attenuated, Double-Deleted Listeria Monocytogenes (pLADD) Immunotherapy in Adults With Metastatic Colorectal Cancer
Brief Title: Study of Personalized Immunotherapy in Adults With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to business realignment
Sponsor: Aduro Biotech, Inc. (Industry)
Collaborators: Hanlee P. Ji, MD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-12
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Neoplasms
Keywords: metastatic; microsatellite stable (MSS)
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): pLADD treatment cycle is once every 3 weeks; starting dose 1×10^8 colony-forming units (CFU) administered IV over 1 hour, and if tolerated increasing to 1×10^9 CFU
  Interventions: Biological: pLADD

INTERVENTIONS:
Biological: pLADD — via IV infusion

SUMMARY:
This study will evaluate the safety and tolerability of a personalized live, attenuated, double-deleted Listeria monocytogenes (pLADD) treatment in adults with metastatic colorectal cancer.

DETAILED DESCRIPTION:
This single arm study is designed to evaluate the safety and tolerability of a personalized treatment in adults with metastatic colorectal cancer by first analyzing the expression of tumor-associated antigens and then treating the patients with a personalized live, attenuated, double-deleted Listeria monocytogenes (pLADD)-based immunotherapy. pLADD is based on the attenuated form of Listeria monocytogenes that has been genetically modified to reduce its ability to cause disease, while maintaining its ability to stimulate a potent immune response. pLADD is manufactured using patient-specific antigens and is therefore individualized to each patient.

ELIGIBILITY:
Inclusion Criteria:

* metastatic colorectal cancer (mCRC) that is microsatellite stable (MSS)
* able to provide adequate tumor tissue from at least 1 accessible tumor site
* completed or have developed intolerance to a course of oxaliplatin- or irinotecan-based frontline therapy at Screening
* on maintenance standard-of-care chemotherapies or on treatment holiday
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* adequate organ function
* progression of disease at the time of Enrollment

Exclusion Criteria:

* BRAF V600E mutation
* known allergy to both penicillin and sulfa drugs
* implanted devices that cannot be easily removed
* immunodeficiency, immune compromised state or receiving immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Through study completion, an average of 12 months
  Number of patients with treatment-related adverse events as assessed by CTCAE v 4.0

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford, Stanford, California
  - Mary Crowley Cancer Research - Medical City, Dallas, Texas